CLINICAL TRIAL: NCT02997007
Title: Investigating the Neural Correlates of Repeated tDCS in MCI and Healthy Ageing With fMRI
Brief Title: Neural Correlates of Repeated tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL57751.068.16
Record Dates: First submitted 2016-11-23; First posted 2016-12-19 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Mild Cognitive Impairment
Keywords: tDCS; Mild Cognitive Impairment; fMRI; Healthy ageing
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MCI-active (Experimental): Patients will receive verum tDCS over the angular gyrus on five consecutive days.
  Interventions: Device: active tDCS
- MCI-sham (Sham Comparator): Patients will receive sham tDCS over the angular gyrus on five consecutive days.
  Interventions: Device: sham tDCS
- Healthy Old-active (Experimental): Participants will receive verum tDCS over the angular gyrus on five consecutive days.
  Interventions: Device: active tDCS
- Healthy old-sham (Sham Comparator): Participants will receive sham tDCS over the angular gyrus on five consecutive days.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — Participants will receive active tDCS over the angular gyrus on five consecutive days
  Arms: Healthy Old-active; MCI-active
Device: sham tDCS — Participants will receive sham tDCS over the angular gyrus on five consecutive days
  Arms: Healthy old-sham; MCI-sham

SUMMARY:
Healthy ageing and pathological ageing in the context of a neurodegenerative disease are both associated with changes in brain network integrity. Episodic memory is especially affected in Alzheimer's disease, but is also decreased in healthy ageing. Consequently, the memory-relevant brain networks are especially altered. Transcranial direct current stimulation (tDCS) has previously been implemented in different clinical- and non-clinical settings and has shown to beneficially influence network connectivity. The neural correlates of single-session tDCS have been investigated, however, the neural effects of repeated tDCS remain unknown. Furthermore, knowledge about the (long-term) neural mechanisms of repeated tDCS can give valuable insights and possibly pave the ground for exploring tDCS as a treatment option in future studies.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Diagnosis of MCI based on the latest research criteria (clinical assessment at the memory clinic (prof. Frans RJ Verhey): presence of at least a memory impairment, memory complaints expressed by the patient or informant, no problems in daily life functioning, no dementia and presence of biomarkers (Albert et al., 2011)
* Clinical Dementia Rating score of 0.5 (CDR distinguishes a stage of questionable dementia (CDR 0.5) from people termed healthy (CDR 0) and those with mild dementia (CDR 1)
* Mini-Mental State Examination (MMSE) 23 and being mentally competent (in general, individuals with a MMSE 18 are considered mentally competent)
* Age: between 60 and 85 years old
* 50% female
* Right-handedness
* Average level of education (CBS level 3-4-5-6)

Healthy controls

* Average neuropsychological test results, in accordance with normative data, corrected for age, education and gender
* No substantial memory complaints (according to the participant)
* Age: between 60 and 85 years old
* 50% female
* Right-handedness
* Average level of education (CBS level 3-4-5-6)
* Normal or corrected to normal vision

Exclusion Criteria:

* Psychoactive medication use
* Abuse of alcohol and drugs
* Cognitive impairment due to alcohol/drug abuse or abuse of other substances
* Past or present psychiatric or neurological disorders (major depression, schizophrenia, bipolar disorder, psychotic disorder (or treatment for it), epilepsy, stroke, Parkinson's disease, multiple sclerosis, brain surgery, brain trauma, electroshock therapy, kidney dialysis, Menière's disease, brain infections)
* Major vascular disorders (e.g. stroke)
* Heart diseases or pacemakers
* Contraindications for scanning (e.g. brain surgery, cardiac pacemaker, metal implants, claustrophobia, body tattoos)
* Large scars or fresh wounds on the scalp

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
neural changes after multi-session tDCS | 5-12 days
  fMRI-BOLD response
network changes after multi-session tDCS | 5-12 days
  functional connectivity between network hubs

SECONDARY OUTCOMES:
Task performance changes after multi-session tDCS | 5-12 days
  BPS-score

CONTACTS AND LOCATIONS:
Overall Officials: Heidi IL Jacobs, PhD, Principal Investigator — Maastricht University; Frans RJ Verhey, Professor, Study Chair — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided